CLINICAL TRIAL: NCT02318134
Title: Fecal Microbiota Transplantation in SAP（Severe Acute Pancreatitis）Patients With Intestinal Barrier Dysfunction
Brief Title: Fecal Microbiota Transplantation for Pancreatitis
Acronym: FMTP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Nanchang University (Other)
Responsible Party: Principal Investigator, Lingyu Luo, Physician-in-charge, The First Affiliated Hospital of Nanchang University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Nanchanguniversity
Record Dates: First submitted 2014-12-12; First posted 2014-12-17 (Estimated); Results first posted 2021-04-14 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-03

CONDITIONS: Acute Pancreatitis; Intestinal Bacteria Flora Disturbance; Intestinal Dysfunction; Fecal Microbiota Transplantation
Keywords: Severe acute pancreatitis; Fecal Microbiota Transplantation; Intestinal barrier dysfunction; Intestinal flora
MeSH Terms: conditions — Pancreatitis | interventions — Fecal Microbiota Transplantation; Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FMT group (Experimental): In the FMT group, participants received 200 mL fresh donor feces for twice (once every two days) via a nasoduodenal tube.
  Interventions: Procedure: Fecal Microbiota Transplantation
- Control group (Placebo Comparator): In the control group, participants received 200 mL normal saline for twice (once every two days) via a nasoduodenal tube.
  Interventions: Drug: normal saline

INTERVENTIONS:
Procedure: Fecal Microbiota Transplantation — FMT via a nasoduodenal tube with fresh bacteria from healthy donor
  Other Names: Fecal Microbiota Therapy; Fecal Transplantation
  Arms: FMT group
Drug: normal saline — Normal saline via a nasoduodenal tube.
  Other Names: normal saline 0.9%
  Arms: Control group

SUMMARY:
The intestinal microbiota plays a pivotal role in the maintenance of intestinal homeostasis and protecting the gut against pathogens by competing for nutrients, creating the intestinal biological barrier and modulating the host immune system.After the onset of acute pancreatitis,the intestinal hypoperfusion and the release of inflammatory mediators result in intestinal barrier dysfunction and intestinal bacteria dysbiosis.This leads to Bacterial and endotoxin translocation, which may cause infectious complications which are major causes of death in SAP patients.Recently,FMT was shown its efficacy in the treatment of gastrointestinal(GI) diseases and non-GI disorders associated with Intestinal flora disturbance by re-establishing the damaged Intestinal Bacteria homeostasis.However,the mechanism by which FMT results in cure of diseases has been poorly understood.This study aims to investigate the therapeutic potential of FMT for SAP patients with intestinal barrier dysfunction.

DETAILED DESCRIPTION:
Investigators aims to restore the intestinal bacteria homeostasis through FMT by retention enema with fresh bacteria,thus stabilizing intestinal barrier dysfunction,minimizing bacterial translocation and preventing infectious complications.The investigators will further examine the effect of FMT on inflammatory markers，the predictors of Intestinal barrier injury and the incidence of infectious complications.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of acute pancreatitis from the First Affiliated Hospital of Nanchang University according to the Classification of acute pancreatitis-2012: revision of the Atlanta classification and definitions by international consensus
2. Onset of pancreatitis within <=2 weeks
3. complicated with gastrointestinal failure. Gastrointestinal failure was defined if the patients were complicated with obvious abdominal distention, abdominal rumbling sound weakening or disappearance, no self-defecation as well as intra-abdominal hypertension.

Exclusion Criteria:

1. SAP complicated by Gastrointestinal bleeding or Intestinal fistula
2. Pregnancy and lactation women
3. Not signed the informed consent
4. Diabetes and autoimmune diseases
5. Multiple organ failure. Organ failure was defined as a score of 2 or more using the modified Marshall scoring system including respiratory failure, renal failure and circulatory.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-11-18 (Actual); Primary Completion 2019-04-17 (Actual); Study Completion 2019-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nonghua Lv, MD, Study Chair — the Frist Affiliated Hospital of Nanchang University
Locations (1):
- the First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi, China

REFERENCES:
- [Background] Liu H, Li W, Wang X, Li J, Yu W. Early gut mucosal dysfunction in patients with acute pancreatitis. Pancreas. 2008 Mar;36(2):192-6. doi: 10.1097/MPA.0b013e31815a399f. PMID 18376312
- [Background] Banks PA, Bollen TL, Dervenis C, Gooszen HG, Johnson CD, Sarr MG, Tsiotos GG, Vege SS; Acute Pancreatitis Classification Working Group. Classification of acute pancreatitis--2012: revision of the Atlanta classification and definitions by international consensus. Gut. 2013 Jan;62(1):102-11. doi: 10.1136/gutjnl-2012-302779. Epub 2012 Oct 25. PMID 23100216
- [Background] Reintam Blaser A, Malbrain ML, Starkopf J, Fruhwald S, Jakob SM, De Waele J, Braun JP, Poeze M, Spies C. Gastrointestinal function in intensive care patients: terminology, definitions and management. Recommendations of the ESICM Working Group on Abdominal Problems. Intensive Care Med. 2012 Mar;38(3):384-94. doi: 10.1007/s00134-011-2459-y. Epub 2012 Feb 7. PMID 22310869
- [Background] Landy J, Al-Hassi HO, McLaughlin SD, Walker AW, Ciclitira PJ, Nicholls RJ, Clark SK, Hart AL. Review article: faecal transplantation therapy for gastrointestinal disease. Aliment Pharmacol Ther. 2011 Aug;34(4):409-15. doi: 10.1111/j.1365-2036.2011.04737.x. Epub 2011 Jun 20. PMID 21682755
- [Background] Smits LP, Bouter KE, de Vos WM, Borody TJ, Nieuwdorp M. Therapeutic potential of fecal microbiota transplantation. Gastroenterology. 2013 Nov;145(5):946-53. doi: 10.1053/j.gastro.2013.08.058. Epub 2013 Sep 7. PMID 24018052
- [Background] Brandt LJ, Aroniadis OC. An overview of fecal microbiota transplantation: techniques, indications, and outcomes. Gastrointest Endosc. 2013 Aug;78(2):240-9. doi: 10.1016/j.gie.2013.03.1329. Epub 2013 May 2. No abstract available. PMID 23642791
- [Background] Seekatz AM, Aas J, Gessert CE, Rubin TA, Saman DM, Bakken JS, Young VB. Recovery of the gut microbiome following fecal microbiota transplantation. mBio. 2014 Jun 17;5(3):e00893-14. doi: 10.1128/mBio.00893-14. PMID 24939885
- [Background] Singh R, Nieuwdorp M, ten Berge IJ, Bemelman FJ, Geerlings SE. The potential beneficial role of faecal microbiota transplantation in diseases other than Clostridium difficile infection. Clin Microbiol Infect. 2014 Nov;20(11):1119-25. doi: 10.1111/1469-0691.12799. Epub 2014 Nov 7. PMID 25274035
- [Background] Allegretti JR, Hamilton MJ. Restoring the gut microbiome for the treatment of inflammatory bowel diseases. World J Gastroenterol. 2014 Apr 7;20(13):3468-74. doi: 10.3748/wjg.v20.i13.3468. PMID 24707129
- [Background] Shankar V, Hamilton MJ, Khoruts A, Kilburn A, Unno T, Paliy O, Sadowsky MJ. Species and genus level resolution analysis of gut microbiota in Clostridium difficile patients following fecal microbiota transplantation. Microbiome. 2014 Apr 21;2:13. doi: 10.1186/2049-2618-2-13. eCollection 2014. PMID 24855561
- [Background] Cui LH, Wang XH, Peng LH, Yu L, Yang YS. [The effects of early enteral nutrition with addition of probiotics on the prognosis of patients suffering from severe acute pancreatitis]. Zhonghua Wei Zhong Bing Ji Jiu Yi Xue. 2013 Apr;25(4):224-8. doi: 10.3760/cma.j.issn.2095-4352.2013.04.011. Chinese. PMID 23660099
- [Derived] Ding L, He C, Li X, Huang X, Lei Y, Ke H, Chen H, Yang Q, Cai Y, Liao Y, He W, Xia L, Xiong H, Lu N, Zhu Y. Efficacy and Safety of Faecal Microbiota Transplantation for Acute Pancreatitis: A Randomised, Controlled Study. Front Med (Lausanne). 2022 Jan 10;8:772454. doi: 10.3389/fmed.2021.772454. eCollection 2021. PMID 35083238
- See also: the First Affiliated Hospital of Nanchang University — http://www.cdyfy.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between November 2017 and April 2019 from the intensive unit care, Department of Gastroenterology, First Affiliated Hospital of Nanchang University.
Period: Overall Study
Arm/Group | FMT Group | Control Group
Started | 30 | 30
Completed | 28 | 29
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FMT Group | Control Group | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.2 (12.4) | 49.9 (13.7) | 48.6 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 12 | 19
  Male | 23 | 18 | 41
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 30 | 30 | 60
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 30 | 30 | 60
BMI [Mean (Standard Deviation); unit: kg/m^2] — Body mass index
  kg/m^2 | 26.3 (3.7) | 25.6 (4.2) | 26.0 (3.9)
Causes of pancreatitis [Count of Participants; unit: Participants]
  Biliary | 9 | 13 | 22
  Alcohol | 6 | 3 | 9
  Hypertriglyceridemia | 14 | 11 | 25
  Other | 1 | 3 | 4
Smoker [Count of Participants; unit: Participants] | 10 | 9 | 19
Drinker [Count of Participants; unit: Participants] | 12 | 8 | 20
Iintra-abdominal pressure [Mean (Standard Deviation); unit: mmHg] | 13.7 (2.4) | 14.5 (2.5) | 14.1 (2.5)
Time from first symptoms to admission [Median (Full Range); unit: days] | 3 [1 to 6] | 3 [1 to 9] | 3 [1 to 9]
Time from admission to intervention [Median (Full Range); unit: days] | 2 [0 to 11] | 1.5 [1 to 8] | 2 [0 to 11]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Gastrointestinal Failure Score Equal 0
Description: The recovery of gastrointestinal dysfunction was assessed by gastrointectinal failure score. Gastrointestinal failure score is a comprehensive score for assessing gastrointestinal function. Gastrointestinal dysfunction score gets o point meaning enteral nutrition> 50% of the required amount and no intra-abdominal hypertension. GIF score range from 0 to 4, and higher scores mean a worse outcome.
Time Frame: one week after intervention
Measure: Count of Participants; unit: Participants
Arm/Group | FMT Group | Control Group
Number analyzed (Participants) | 30 | 30
Participants | 12 | 14

2. Secondary Outcome: Number of Participants With Infectious Complications
Description: The incidence of any infectious complications，such as infected pancreatic necrosis, infected ascites, bacteraemia, pneumonia, urinary tract infection.
Time Frame: 120 days
Measure: Count of Participants; unit: Participants
Arm/Group | FMT Group | Control Group
Number analyzed (Participants) | 30 | 30
Participants
  Any infectious complications | 15 | 16
  Documented IPN | 4 | 8
  Suspected or documented IPN | 10 | 9
  infected ascites | 2 | 2
  bacteremia | 9 | 10
  pneumonia | 6 | 8
  Urinary tract infection | 3 | 7

3. Secondary Outcome: Number of Participants With Organ Failure
Description: The incidence of organ failure,such as respiratory failure, renal failure, circulatory failure.
Time Frame: 120 days
Measure: Count of Participants; unit: Participants
Arm/Group | FMT Group | Control Group
Number analyzed (Participants) | 30 | 30
Participants
  Any persistent organ failure | 24 | 23
  Persistent respiratory failure | 24 | 21
  Persistent renal failure | 3 | 5
  Persistent circulatory failure | 9 | 11

4. Secondary Outcome: Number of Participants With Interventions or Surgery
Description: number of patients who need extra interventions or surgery
Time Frame: 120 days
Measure: Count of Participants; unit: Participants
Arm/Group | FMT Group | Control Group
Number analyzed (Participants) | 30 | 30
Participants
  Percutaneous or endoscopic transmural drainage | 10 | 11
  Percutaneous or endoscopic transmural necrosectomy | 6 | 7
  Open surgery | 1 | 1
  Mechanical ventilation | 12 | 10
  Renal replacement therapy | 2 | 3

5. Secondary Outcome: Length of Intensive Care Time and Hospital Stay
Description: patients' Length of Intensive care time and hospital stay due to the disease
Time Frame: 6 months
Measure: Median (Full Range); unit: days
Arm/Group | FMT Group | Control Group
Number analyzed (Participants) | 30 | 30
days
  Intensive care stay | 9 [3 to 103] | 11 [2 to 43]
  Hospital stay | 18.5 [9 to 122] | 23 [5 to 125]

6. Secondary Outcome: Mortality
Description: patients who die due to the diseases
Time Frame: 120 days
Measure: Count of Participants; unit: Participants
Arm/Group | FMT Group | Control Group
Number analyzed (Participants) | 30 | 30
Participants | 3 | 4

7. Secondary Outcome: Diamine Oxidase（DAO）
Description: Plasma Diamine oxidase（DAO）level as a predictor in the diagnosis of Intestinal mucosal barrier injury. The rate of decline in DAO was calculated by ((value before intervention - value one week after intervention)/ value before intervention)*100)
Time Frame: one week after intervention
Measure: Median (Full Range); unit: percent change of DAO
Arm/Group | FMT Group | Control Group
Number analyzed (Participants) | 30 | 30
percent change of DAO | -0.21 [-46.2 to 0.57] | -0.05 [-4.32 to 0.78]

8. Secondary Outcome: D-lactate
Description: Plasma D-lactate level as a predictor in the diagnosis of Intestinal mucosal. The rate of decline in D-lactate was calculated by ((value before intervention - value one week after intervention)/ value before intervention)*100).
Time Frame: one week after intervention
Measure: Median (Full Range); unit: percent change of D-lactate
Arm/Group | Control Group | FMT Group
Number analyzed (Participants) | 30 | 30
percent change of D-lactate | 0.37 [-1.06 to 0.85] | -0.28 [-3.72 to 0.75]

ADVERSE EVENTS:
Time Frame: 10 months
Arm/Group | FMT Group | Control Group
All-Cause Mortality (participants affected / at risk) | 3/30 | 4/30
Serious Adverse Events (participants affected / at risk) | 24/30 | 24/30
Other Adverse Events (participants affected / at risk) | 25/30 | 25/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FMT Group (N=30) | Control Group (N=30)
Infected pancreatic necrosis (Infections and infestations) | 4 (4) | 8 (8) — Positive culture of peripancreatic fluid or pancreatic necrosis obtained by either fine-needle aspiration or during the first percutaneous or endoscopic drainage
Persistent respiratory failure (Respiratory, thoracic and mediastinal disorders) | 24 (24) | 21 (21) — PaO2/FiO2 below 300
Persistent renal failure (Renal and urinary disorders) | 3 (3) | 5 (5) — Serum Creatinine over 170 μmol/l or 1.9 mg/dl
Persistent circulatory failure (Cardiac disorders) | 9 (9) | 11 (11) — Systolic blood pressure below 90 mm Hg, not fluid responsive or pH below 7.3
gastrointestinal fistula (Gastrointestinal disorders) | 1 (1) | 1 (1)
intra-abdominal bleeding (Gastrointestinal disorders) | 2 (2) | 0 (0)
gastrointestinal bleeding (Gastrointestinal disorders) | 2 (2) | 1 (1)
gastrointestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FMT Group (N=30) | Control Group (N=30)
infected ascites (Infections and infestations) | 2 (2) | 2 (2) — bacteria or fungi detected in aspirate of intraperitoneal fluid
Bacteraemia (Infections and infestations) | 9 (9) | 10 (10) — positive blood culture
pneumonia (Infections and infestations) | 6 (6) | 8 (8) — Positive sputum or endotracheal culture
Urinary tract infection (Infections and infestations) | 3 (3) | 7 (7) — Positive urine culture
bloating (Gastrointestinal disorders) | 25 (25) | 24 (24)
vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-15): https://cdn.clinicaltrials.gov/large-docs/34/NCT02318134/Prot_SAP_000.pdf